CLINICAL TRIAL: NCT00344331
Title: Evaluation of Biochemical Markers and Clinical Investigation of Niemann-Pick Disease, Type C
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060186; 06-CH-0186
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-10-01

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Lysosomal Storage; Biomarkers; Longitudinal; Natural History; Niemann Pick Type C; NPC; Lysosomal Storage Disorder
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Volunteers may be of varying age, with no contraindication to collection of biospecimen.
- Patients with a diagnosis of Niemann-Pick type C (NPC) of either sex and any age: Participants may range from neurologically asymptomatic to severe and may have liver disease or unrelated comorbidities, but must be stable enough to safely travel and tolerate medical evaluations.

SUMMARY:
This study will evaluate clinical and laboratory tests that might be useful in determining if an investigational drug can slow the progression of Niemann-Pick Disease, Type C (NPC), a genetic disorder that results in progressive loss of nervous system function. The study will: 1) look for a clinical or biochemical marker that can be used as a measure of response to treatment, and 2) define the rate of progression of biochemical marker abnormalities in a group of NPC patients who will later be invited to enroll in a treatment trial.

Patients of any age with NPC may be eligible for this study. Participants undergo the following procedures every 6 months during 4- to 5-day admissions at the NIH Clinical Center.

* Medical evaluation, including medical history, physical exam, neurological exam, neuropsychometric evaluation, and blood and urine tests.
* Lumbar puncture (spinal tap): A sample of cerebrospinal fluid (CSF), the fluid that bathes the brain and spinal cord, is obtained for study. After administration of a local anesthetic, a small needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. A small amount of fluid is collected through the needle.
* Eye exam and eye movement study: The pupils of the eye are dilated to examine the structures of the eyes. For the eye movement study a special contact lens is placed on the eye and the patient looks at a series of target light spots moving on a screen.
* Hearing tests.
* Electroretinography (in patients who can cooperate with the test) to measure the function of the retina. Before the test, the patient's pupils are dilated and an electrode (small silver disk) is taped to the forehead. The patient sits in a dark room for 30 minutes and then a special contact lens is placed on one eye after it has been numbed with drops. The contact lens senses small electrical signals generated by the retina when lights flash. During the ERG recording, the eye is stimulated with flashes of light projected inside a hollow sphere. After the test, a full eye exam is done and photographs of the retina are taken.
* Magnetic resonance imaging (MRI): This test uses a magnetic field and radio waves to produce images of the brain and obtain information about brain chemicals. The patient lies on a table that can slide in and out of the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. Patients who cannot remain still in the scanner may be sedated for the test.
* Psychometric testing: Patients complete questionnaires.
* Photographs of the patient may be taken for use in teaching sessions or scientific presentations or publications, with the patient's consent. Patients may be recognizable, but are not identified by name.
* Pregnancy test in all female patients over 10 years of age at the beginning of each admission to the Clinical Center.

DETAILED DESCRIPTION:
Niemann-Pick type C disease (NPC) is an autosomal recessive, lysosomal storage disorder characterized by accumulation of cholesterol and gangliosides. NPC is a rare (estimated prevalence of 1:120,000-150,000) neurodegenerative disorder with a wide clinical spectrum and a variable age of onset. Classically, children with NPC demonstrate neurological dysfunction with cerebellar ataxia, dysarthria, seizures, vertical gaze palsy, motor impairment, dysphagia, psychotic episodes, and progressive dementia. In general, adolescent and adult onset forms have a more insidious onset and slower progression.

There is no effective treatment for NPC and it is a lethal disorder. A major impediment to the testing of therapeutic interventions is the lack of well-defined outcome measures. The purpose of this protocol is to obtain both baseline and rate of progression data on clinical and biochemical markers that may later be used as an outcome measure in a clinical trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected Subjects

The following individuals may be enrolled as in this study:

* All patients with a diagnosis of NPC, based on clinical presentation, biochemical, or molecular.
* Both NPC1 and NPC2 patients.
* Patients of any age
* Males or females
* Any ethnic background

EXCLUSION CRITERIA:

Individuals will not be enrolled in this study if:

* they cannot travel to the NIH because of their medical condition or are too ill to be cared for at home.
* they have rapidly progressive neonatal cholestasis.
* they are pregnant (a negative urine pregnancy test will be required for any menstruating female before participation in this study and at each NIH Clinical Center admission).

Unaffected Subjects

Individuals may be enrolled for data and biospecimen collection if:

* They are a known NPC1 or NPC2 heterozygote and consent to specimen collection (as specified in the protocol) from the carrier population.
* There is no diagnosis or suspicion of NPC disease, and consent is provided to be included in control or caregiver population.

Individuals will not be enrolled for biospecimen collection if:

* Consent is not provided
* They have a contraindication to the method of specimen collection

  * Patients will be excluded from the MRI section of the study if they have a contraindication to MRI or if they do not meet the safety criteria established by the NIH Clinical Center radiology department for MRI scanning.

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age with Niemann-Pick type C
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2006-08-14 (Actual)

PRIMARY OUTCOMES:
Plasma Oxysterols | Ad Hoc
  Oxysterols such as 24S-hydroxycholesterol, 25-hydroxycholesterol, and 27-hydroxycholesterol are derived from cholesterol and play a role in cholesterol homeostasis. No data is available on endogenous oxysterol levels in NPC patients. We plan to measure oxysterol levels in both serum and CSF and correlate these levels with disease status and progression.
Clinical & Biochemical Markers | Ad Hoc
  Identify a clinical and/or biochemical marker that can be used as a therapeutic outcome measure for NPC.
Define Rate of Progression | Ad Hoc
  Define rate of progression of biochemical marker abnormalities in <TAB>NPC patients for future therapeutic indication.

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will be coded and shared in aggregate.

REFERENCES:
- [Background] Solomon BI, Smith AC, Sinaii N, Farhat N, King MC, Machielse L, Porter FD. Association of Miglustat With Swallowing Outcomes in Niemann-Pick Disease, Type C1. JAMA Neurol. 2020 Dec 1;77(12):1564-1568. doi: 10.1001/jamaneurol.2020.3241. PMID 32897301
- [Derived] Farmer C, Lewis M, Farhat N, Robbins KP, Joseph L, Albert OK, Bianconi S, Hoffmann A, Giserman-Kiss I, Alexander DM, Thurm A, Porter FD, Kravis EB. Convergent Validity of the Fine Motor, Speech, and Cognitive Domains of the 5-Domain Niemann-Pick Disease Type C Clinical Severity Scale. J Child Neurol. 2026 Jan;41(1):43-53. doi: 10.1177/08830738251346348. Epub 2025 Jun 17. PMID 40525490
- [Derived] Campbell K, Cawley NX, Luke R, Scott KEJ, Johnson N, Farhat NY, Alexander D, Wassif CA, Li W, Cologna SM, Berry-Kravis E, Do AD, Dale RK, Porter FD. Identification of cerebral spinal fluid protein biomarkers in Niemann-Pick disease, type C1. Biomark Res. 2023 Jan 31;11(1):14. doi: 10.1186/s40364-023-00448-x. PMID 36721240
- [Derived] Solomon BI, Munoz AM, Sinaii N, Farhat NM, Smith AC, Bianconi S, Dang Do A, Backman MC, Machielse L, Porter FD. Phenotypic expression of swallowing function in Niemann-Pick disease type C1. Orphanet J Rare Dis. 2022 Sep 5;17(1):342. doi: 10.1186/s13023-022-02472-w. PMID 36064725
- [Derived] Thurm A, Chlebowski C, Joseph L, Farmer C, Adedipe D, Weiss M, Wiggs E, Farhat N, Bianconi S, Berry-Kravis E, Porter FD. Neurodevelopmental Characterization of Young Children Diagnosed with Niemann-Pick Disease, Type C1. J Dev Behav Pediatr. 2020 Jun/Jul;41(5):388-396. doi: 10.1097/DBP.0000000000000785. PMID 32073546
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2006-CH-0186.html